CLINICAL TRIAL: NCT00716183
Title: Phase 2/3 Evaluation of Three Lactobacilli Strains Isolated From Human Milk for the Treatment of Infectious Mastitis During the Lactation Period
Brief Title: Use of Probiotic Lactobacilli for the Treatment of Lactational Mastitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Juan M. Rodríguez, Universidad Complutense de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Promast08
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Mastitis
Keywords: mastitis; Staphylococcus; Streptococcus; lactation; breastfeeding
MeSH Terms: conditions — Mastitis; Breast Feeding | interventions — Monobactams; Amoxicillin; Drugs, Generic; Cloxacillin; Clavulanic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Probiotic 1 (Experimental): Women receiving Lactobacillus salivarius HN6
  Interventions: Biological: Lactobacillus salivarius HN6
- Probiotic 2 (Experimental): Women receiving Lactobacillus reuteri CR20
  Interventions: Biological: Lactobacillus reuteri CR20
- Probiotic 3 (Experimental): Women receiving Lactobacillus fermentum LC40
  Interventions: Biological: Lactobacillus fermentum LC40
- beta-lactam (Active Comparator): The evolution of the women ascribed to the other three arms will be compared with that of 100 women suffering lactational mastitis that will follow a conventional antibiotic treatment as prescribed by the pediatrician/gynecologist
  Interventions: Drug: Beta-lactam antibiotic

INTERVENTIONS:
Biological: Lactobacillus salivarius HN6 — 9 log colony-forming units, capsules, daily, four weeks
  Arms: Probiotic 1
Biological: Lactobacillus reuteri CR20 — 9 log colony-forming units, capsules, daily, four weeks
  Arms: Probiotic 2
Biological: Lactobacillus fermentum LC40 — 9 log colony-forming units, capsules, daily, four weeks
  Arms: Probiotic 3
Drug: Beta-lactam antibiotic — Use of amoxicillin, cloxacillin or amoxicillin/clavulanic acid(500-750 mg), orally, every 8-12 h, for 2-3 weeks (as prescribed by the physician responsible for the clinical diagnosis of lactational mastitis)
  Other Names: Amoxicillin (generic), Cloxacillin (generic), Amoxicillin/clavulanic acid (generic), Clamoxyl, Orbenin, Augmentine
  Arms: beta-lactam

SUMMARY:
A total of 300 women with lactational infectious mastitis will daily ingest 9 log10 cfu of Lactobacillus salivarius HN6, Lactobacillus reuteri CR20 or Lactobacillus fermentum LC40 for 4 weeks. The three lactobacilli strains were originally isolated from milk of healthy women. On days 0 and 28, milk samples will be collected, and staphylococci/streptococci and lactobacilli will be counted and identified. Evolution of clinical signs will be recorded by midwifes on days 0, 7, 14 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mastitis
* Staphylococcal and/or streptococcal count higher than 3000 colony-forming units per ml of milk
* Milk leukocyte count higher 6 log10/mL
* Must be able to provide a milk sample without the aid of a milk pump

Exclusion Criteria:

* Mammary abscesses
* Any kind of parallel disease

Ages: 19 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Staphylococcal and/or streptococcal count in milk | 0 and 28 days

SECONDARY OUTCOMES:
Assessment of local and systemic symptoms associated to mastitis | days 0, 7, 14 and 28

CONTACTS AND LOCATIONS:
Locations (1):
- Dpt. Nutricion, Bromatologia y Tecnologia de los Alimentos, Madrid, Madrid, Spain

REFERENCES:
- [Background] Jimenez E, Fernandez L, Maldonado A, Martin R, Olivares M, Xaus J, Rodriguez JM. Oral administration of Lactobacillus strains isolated from breast milk as an alternative for the treatment of infectious mastitis during lactation. Appl Environ Microbiol. 2008 Aug;74(15):4650-5. doi: 10.1128/AEM.02599-07. Epub 2008 Jun 6. PMID 18539795
- [Background] Martin R, Olivares M, Marin ML, Fernandez L, Xaus J, Rodriguez JM. Probiotic potential of 3 Lactobacilli strains isolated from breast milk. J Hum Lact. 2005 Feb;21(1):8-17; quiz 18-21, 41. doi: 10.1177/0890334404272393. PMID 15681631
- [Background] Martin R, Langa S, Reviriego C, Jiminez E, Marin ML, Xaus J, Fernandez L, Rodriguez JM. Human milk is a source of lactic acid bacteria for the infant gut. J Pediatr. 2003 Dec;143(6):754-8. doi: 10.1016/j.jpeds.2003.09.028. PMID 14657823
- [Background] Martin R, Heilig GH, Zoetendal EG, Smidt H, Rodriguez JM. Diversity of the Lactobacillus group in breast milk and vagina of healthy women and potential role in the colonization of the infant gut. J Appl Microbiol. 2007 Dec;103(6):2638-44. doi: 10.1111/j.1365-2672.2007.03497.x. PMID 18045446
- [Background] Delgado S, Arroyo R, Martin R, Rodriguez JM. PCR-DGGE assessment of the bacterial diversity of breast milk in women with lactational infectious mastitis. BMC Infect Dis. 2008 Apr 18;8:51. doi: 10.1186/1471-2334-8-51. PMID 18423017
- [Background] Martin R, Jimenez E, Olivares M, Marin ML, Fernandez L, Xaus J, Rodriguez JM. Lactobacillus salivarius CECT 5713, a potential probiotic strain isolated from infant feces and breast milk of a mother-child pair. Int J Food Microbiol. 2006 Oct 15;112(1):35-43. doi: 10.1016/j.ijfoodmicro.2006.06.011. Epub 2006 Jul 14. PMID 16843562
- [Background] Olivares M, Diaz-Ropero MP, Martin R, Rodriguez JM, Xaus J. Antimicrobial potential of four Lactobacillus strains isolated from breast milk. J Appl Microbiol. 2006 Jul;101(1):72-9. doi: 10.1111/j.1365-2672.2006.02981.x. PMID 16834593
- [Derived] Vazquez-Fresno R, Llorach R, Marinic J, Tulipani S, Garcia-Aloy M, Espinosa-Martos I, Jimenez E, Rodriguez JM, Andres-Lacueva C. Urinary metabolomic fingerprinting after consumption of a probiotic strain in women with mastitis. Pharmacol Res. 2014 Sep;87:160-5. doi: 10.1016/j.phrs.2014.05.010. Epub 2014 May 29. PMID 24880136
- [Derived] Arroyo R, Martin V, Maldonado A, Jimenez E, Fernandez L, Rodriguez JM. Treatment of infectious mastitis during lactation: antibiotics versus oral administration of Lactobacilli isolated from breast milk. Clin Infect Dis. 2010 Jun 15;50(12):1551-8. doi: 10.1086/652763. PMID 20455694